CLINICAL TRIAL: NCT03401372
Title: Comparison of Bortezomib-Cyclophosphamide-Dexamethasone Chemotherapy With or Without Doxycycline in Newly Diagnosed Mayo Stage II-III Light Chain Amyloidosis Patients: A Multi-center Randomized Controlled Trial
Brief Title: BCD With or Without Doxycycline in Mayo Stage II-III Light Chain Amyloidosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jian Li (Other)
Collaborators: Peking University First Hospital (Other); Beijing Anzhen Hospital (Other); Beijing Chao Yang Hospital (Other); West China Hospital (Other); Tongji Hospital (Other); Union Hospital Affiliated with Tongji Medical College of HUST (Unknown); Shanghai Changzheng Hospital (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor-Investigator, Jian Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-AL2017
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Amyloidosis; Systemic
Keywords: Primary light chain amyloidosis; Doxycycline; Bortezomib; Prognosis; Progression-free survival; Overall survival; Organ response
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Doxycycline; Bortezomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycycline/BCD chemotherapy (Experimental): Doxycycline combined with bortezomib-cyclophosphamide-dexamethasone chemotherapy
  Interventions: Drug: Doxycycline; Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Dexamethasone
- BCD chemotherapy (Active Comparator): Bortezomib-cyclophosphamide-dexamethasone chemotherapy
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Doxycycline — Oral doxycycline 100mg twice daily
  Arms: Doxycycline/BCD chemotherapy
Drug: Bortezomib — 1.3mg/m2 of bortezomib on days 1, 8, 15 and 22 of a 35-day cycle
Drug: Cyclophosphamide — 300mg/m2 cyclophosphamide on days 1, 8, 15 and 22 of a 35-day cycle
Drug: Dexamethasone — 40mg of dexamethasone on days 1, 8, 15 and 22 of a 35-day cycle

SUMMARY:
Survival of intermediate and high-risk primary light chain amyloidosis (pAL) remains poor due to high mortality within 3-6 months of diagnosis. Rapidly effective regimens such as bortezomib, cyclophosphamide and dexamethasone (BCD) still failed to overcome the poor prognosis in very advanced pAL amyloidosis patients. Recently, doxycycline was demonstrated to induce disruption of fibril formation and reduce the number of intact fibrils in transgenic mouse model of pAL amyloidosis. Furthermore, case-control study suggested that adjuvant oral doxycycline could improve response and survival in cardiac pAL amyloidosis, which necessities further confirmation through a randomized trial. Therefore, we designed a multi-center randomized open-label controlled study to investigate the efficacy and safety of co-administration of oral doxycycline with BCD regimen in treatment-naïve patients with Mayo stage II-III pAL amyloidosis. The primary outcome progression-free survival, and secondary endpoints including overall survival, hematologic response, organ response and toxicity of doxycycline will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old adults.
* Biopsy proved treatment-naïve pAL amyloidosis.
* Mayo 2004 stage II-III.
* dFLC > 50mg/L.
* Patient must provide informed consent.

Exclusion Criteria:

* Co-morbidity of uncontrolled infection.
* Co-morbidity of grade 2 or 3 atrioventricular block.
* Co-morbidity of sustained or recurrent nonsustained ventricular tachycardia.
* Co-morbidity of other active malignancy.
* Co-diagnosis of multiple myeloma or waldenstrom macroglobulinemia.
* Grade 2 or higher neuropathy according to National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0.
* Allergic history of doxycycline.
* Neutrophil <1×10E9/L，hemoglobin < 7g/dL，or platelet < 75×10E9/L.
* Severely compromised hepatic or renal function: ALT or AST > 2.5 × ULN, total bilirubin > 1.5mg/dL，or eGFR < 60mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  The patients are assessed after each cycle of chemotherapy following treatment initiation until progression, relapse, death or study closure at 24-month follow-up.

SECONDARY OUTCOMES:
Overall survival | 2 years
  The patients are assessed after each cycle of chemotherapy following treatment initiation until progression, relapse, death or study closure at 24-month follow-up. If the primary endpoint has reached, patients will also be followed up every 3 months thereafter until death or study closure.
Hematologic response | 2 years
  The patients are assessed after each cycle of chemotherapy following treatment initiation until progression, relapse, death or study closure at 24-month follow-up. If the primary endpoint has reached, patients will also be followed up every 3 months thereafter until death or study closure.
Organ response | 2 years
  The patients are assessed after each cycle of chemotherapy following treatment initiation until progression, relapse, death or study closure at 24-month follow-up. If the primary endpoint has reached, patients will also be followed up every 3 months thereafter until death or study closure.
Adverse events | up to 2 years
  Adverse events are collected until 30 days after last dose of doxycycline.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ward JE, Ren R, Toraldo G, Soohoo P, Guan J, O'Hara C, Jasuja R, Trinkaus-Randall V, Liao R, Connors LH, Seldin DC. Doxycycline reduces fibril formation in a transgenic mouse model of AL amyloidosis. Blood. 2011 Dec 15;118(25):6610-7. doi: 10.1182/blood-2011-04-351643. Epub 2011 Oct 12. PMID 21998211
- [Result] Shen KN, Li J. [Light Chain Amyloidosis: an Update for Treatment]. Zhongguo Shi Yan Xue Ye Xue Za Zhi. 2015 Jun;23(3):910-4. doi: 10.7534/j.issn.1009-2137.2015.03.059. Chinese. PMID 26117060
- [Result] Feng J, Huang XF, Zhang CL, Shen KN, Zhang CL, Sun J, Tian Z, Cao XX, Zhang L, Zhou DB, Li J. [Analysis of clinical characteristics and outcome of patients with very high risk primary immunoglobulin light-chain amyloidosis]. Zhonghua Xue Ye Xue Za Zhi. 2017 Feb 14;38(2):107-111. doi: 10.3760/cma.j.issn.0253-2727.2017.02.005. Chinese. PMID 28279033
- [Result] Dispenzieri A, Gertz MA, Kyle RA, Lacy MQ, Burritt MF, Therneau TM, Greipp PR, Witzig TE, Lust JA, Rajkumar SV, Fonseca R, Zeldenrust SR, McGregor CG, Jaffe AS. Serum cardiac troponins and N-terminal pro-brain natriuretic peptide: a staging system for primary systemic amyloidosis. J Clin Oncol. 2004 Sep 15;22(18):3751-7. doi: 10.1200/JCO.2004.03.029. PMID 15365071
- [Result] Mikhael JR, Schuster SR, Jimenez-Zepeda VH, Bello N, Spong J, Reeder CB, Stewart AK, Bergsagel PL, Fonseca R. Cyclophosphamide-bortezomib-dexamethasone (CyBorD) produces rapid and complete hematologic response in patients with AL amyloidosis. Blood. 2012 May 10;119(19):4391-4. doi: 10.1182/blood-2011-11-390930. Epub 2012 Feb 13. PMID 22331188
- [Result] Venner CP, Gillmore JD, Sachchithanantham S, Mahmood S, Lane T, Foard D, Rannigan L, Gibbs SD, Pinney JH, Whelan CJ, Lachmann HJ, Hawkins PN, Wechalekar AD. A matched comparison of cyclophosphamide, bortezomib and dexamethasone (CVD) versus risk-adapted cyclophosphamide, thalidomide and dexamethasone (CTD) in AL amyloidosis. Leukemia. 2014 Dec;28(12):2304-10. doi: 10.1038/leu.2014.218. Epub 2014 Jul 16. PMID 25027514
- [Result] Kastritis E, Roussou M, Gavriatopoulou M, Migkou M, Kalapanida D, Pamboucas C, Kaldara E, Ntalianis A, Psimenou E, Toumanidis ST, Tasidou A, Terpos E, Dimopoulos MA. Long-term outcomes of primary systemic light chain (AL) amyloidosis in patients treated upfront with bortezomib or lenalidomide and the importance of risk adapted strategies. Am J Hematol. 2015 Apr;90(4):E60-5. doi: 10.1002/ajh.23936. Epub 2015 Mar 9. PMID 25580702
- [Derived] Shen KN, Fu WJ, Wu Y, Dong YJ, Huang ZX, Wei YQ, Li CR, Sun CY, Chen Y, Miao HL, Zhang YL, Cao XX, Zhou DB, Li J. Doxycycline Combined With Bortezomib-Cyclophosphamide-Dexamethasone Chemotherapy for Newly Diagnosed Cardiac Light-Chain Amyloidosis: A Multicenter Randomized Controlled Trial. Circulation. 2022 Jan 4;145(1):8-17. doi: 10.1161/CIRCULATIONAHA.121.055953. Epub 2021 Sep 10. PMID 34503349